CLINICAL TRIAL: NCT02721719
Title: The Role of CD4+ T Cell Subsets in the Mechanism of Action of Vedolizumab in Ulcerative Colitis
Status: Active, not recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Brian Bressler, Clinical Assistant Professor, University of British Columbia
Other Study IDs: H15-01034
Record Dates: First submitted 2016-03-08; First posted 2016-03-29 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; UC; Vedolizumab; Entyvio; Inflammatory Bowl Disease; IBD; T-Lymphocytes, Regulatory
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood & colonic biopsy tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy Adults: [Not receiving Vedolizumab] Healthy adults who have not donated blood within the past two months and who have no history of blood-borne diseases.
- Adults with no Inflammatory Bowl Disease: [Not receiving Vedolizumab] Adult patients undergoing endoscopy for indications other than Inflammatory Bowel Disease or other inflammatory conditions of the bowel (such as colon cancer screening or polypectomy)
- Donors with Ulcerative Colitis: [Set to receive Vedolizumab] Adults with an established diagnosis of UC (≥ 6 months preceding involvement in study) who are both scheduled for an endoscopy and are about to receive Vedolizumab treatment (standard of care).

SUMMARY:
The cause of Inflammatory Bowl Disease (IBD) is not known, but studies from patients with IBD have found that these patients make unusually strong immune responses to their own intestinal tissues and to bacteria that normally live in the healthy gut. These overactive immune responses might result from an imbalance of T-lymphocytes, which are a type of white blood cell that recognize and respond to threats like infection or damaged tissues. In healthy tissues, a type of T-lymphocytes called T-regulatory cells control excess inflammation by preventing other T cells, called T-effector cells from responding. We believe that T-regulatory cells are somehow less active in IBD, resulting in damage to intestinal tissues by the T-effector cells.

T-lymphocytes, including both T-regulatory and T-effector cells, are guided to different parts of the body by 'alpha4beta7-integrin' molecules. Vedolizumab or Entyvio works by blocking this homing molecule so that T cells do not reach the intestine, but stay in the blood where they cannot aggravate your IBD. This study will help in understanding how Vedolizumab helps to heal or decrease the symptoms of your Ulcerative Colitis.

The effect of Vedolizumab on different types of T cells in the human intestine has not yet been studied. However, the investigators think that Vedolizumab will shift the balance of T cells in the intestine towards more healing T-regulatory cells and less damaging T-effector cells. The purpose of this study is to measure the different types of T cells in participants' blood and intestinal tissue before and during Vedolizumab treatment.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is an umbrella term for Crohn's disease and Ulcerative Colitis (UC), which are thought to be caused by disruption of the intestinal epithelial cell barrier, leading to changes in the intestinal flora and a consequent aberrant activation of the mucosal immune system. The resulting chronic intestinal inflammation is highly dependent on different subsets of CD4+ T helper (Th) cells. For example, correlative data suggest that Crohn's disease is driven by exaggerated Th1 and Th17 cell responses, since inflamed lesions contain increased levels of cytokines associated with these cells including IFNγ, IL-12, and IL-17 and IL-18. In contrast, although Ulcerative Colitis is in the same family of diseases, it is typically associated with Th2 cells since patients have high levels of IL-13 in the intestinal mucosa compared to patients with Crohn's disease or healthy individuals. Recent evidence implicates the newly emerging Th9 subset of Th cells in the pathology of UC. The development and function of Th cells with pathogenic potential is kept in check by another subset of CD4+ T cells, which is known as the regulatory T cell, or Treg. In healthy individuals, the intestinal lamina propria has a large proportion of Tregs, and evidence that simply lacking Tregs leads to IBD, suggests Tregs have a critical role in controlling intestinal homeostasis. Indeed, work in animal models and early phase clinical trials have shown that restoration of Treg function can ameliorate IBD. These data suggest that effective therapies need to promote the function of Tregs. Hence in order to understand the mechanism of action of new therapeutics it is critical to assess their impact on the balance between effector and regulatory CD4+ T cells.

Homing of effector and regulatory T cells to the intestine is controlled by a variety of integrins and chemokine receptors, with evidence that expression of alpha4beta7-integrin molecules (α4β7) on T cells has a key role in this process. Since Vedolizumab (Entyvio) specifically blocks the interaction between α4β7 and its ligands, which are expressed in mucosal tissue, its therapeutic effects in IBD are presumed to be related to a reduction in T cell trafficking to the intestine. However, how this biologic agent specifically affects the homing of Tregs versus effector T cells is unknown. In humans, Tregs in the peripheral blood are reported to express lower levels of α4β7 compared to effector T cells, but the relative expression on different subsets (i.e. Th1, vs. Th2, vs. Th17) of CD4+ T cells is unknown. Interestingly, in the intestine there is also a subset of Tregs that produces IL-17 and expresses high levels of α4β7, but the functional relevance of these cells in IBD is unknown. In addition, in mice, expression of α4β7 on CD4+ T cells is unstable under inflammatory conditions, suggesting that studies with circulating T cells in healthy individuals may not accurately reflect integrin expression in states of inflammation. Understanding how Vedolizumab affects the localization of circulating versus tissue-localized subsets of CD4+ T cells is key to understanding how this therapy works.

Also unknown is how signaling by α4β7 affects the development and/or function of different subsets of CD4+ T cells. In T cells, integrins not only mediate homing, but they also provide tissue-specific signals. For example, they can act as costimulatory molecules 10-12 and influence cytokine production. The molecular basis for the effects on T cells has not been well characterized, but in other cells integrins activate the PI3K pathway, providing a pro-survival signal 16. Since we have shown that activation of the PI3K pathway regulates the balance of effector versus regulatory T cells 17, it is possible that blockade of α4β7 may reduce PI3K signaling and favor the development of Tregs. In support of this possibility, we have shown that fibronectin, which is a ligand for α4β7, inhibits the development of Tregs.

This is an observational study to determine the expression pattern and function of α4β7 on effector and regulatory CD4+ T cells, and to define how treatment with Vedolizumab affects the homing and function of these cells. We hypothesize that that treatment with Vedolizumab will shift the balance of effector and regulatory T cells through two mechanisms: 1) altered migration of different subsets of CD4+ T cells to the intestine; and 2) promoting Treg stability as a consequence of reduced PI3K signaling downstream of α4β7.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Healthy adults who have not donated blood within the past two months and who have no history of blood-borne diseases.
* Group 2: Adult patients undergoing endoscopy for indications other than Inflammatory Bowel Disease or other inflammatory conditions of the bowel (such as colon cancer screening or polypectomy)
* Group 3: Adults with an established diagnosis of Ulcerative Colitis (≥ 6 months preceding involvement in study) who are both scheduled for an endoscopy and are about to receive Vedolizumab as part of their standard of care treatment. Former anti-TNF treated Ulcerative Colitis patients will not be excluded, however, only 50% of the group 3 patient cohort can be on anti-TNF medications 12 weeks before Vedolizumab initiation.

Exclusion Criteria:

* Less than 19 years of age or greater than 80 years of age
* Known or suspected inflammatory conditions of the bowel (such as irritable bowel syndrome, celiac disease)
* Known or suspected transmissible infectious disease such as HIV, Hep B or C or a hemorrhagic disorder
* Known hematologic malignancy
* Pregnancy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Healthy human volunteers who respond to our advertising poster (put up around CFRI and Vancouver General Hospital).
  Group 2: Patients who are undergoing endoscopy at the Pacific Gastroenterology Associate's endoscopy clinic for indications other than Inflammatory Bowel Disease (such as colon cancer screening or polypectomy).
  Group 3: Participants who are about to undergo Vedolizumab treatment from Pacific Gastroenterology Associate's clinic (affiliated with St. Paul's Hospital) as part of their standard of care treatment. Physicians will identify these patients when they undergo medical consultation for treatment of their Ulcerative Colitis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-05; Primary Completion 2023-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Differences in CD4+ T cell subsets in the blood and colonic tissue of IBD patients before and after Vedolizumab treatment; relative CD4+ T cell numbers will be determined by immunofluorescent detection of subset specific markers. | Two years

SECONDARY OUTCOMES:
Differences in the stability of T regulatory cells with and without alpha4beta7 integrin binding as measured by maintenance of the Treg-specific-demethylation region in the FoxP3 promoter. | Two years
Differences in the suppressive capacity of T regulatory cells with and without alpha4beta7 integrin binding as measured by ability to suppress the proliferation of CD4+CD25- T effector cells. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Brian Bressler, MD, FCRP(C), Principal Investigator — University of British Columbia
Locations (1):
- Child and Family Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardenberg G, Steiner TS, Levings MK. Environmental influences on T regulatory cells in inflammatory bowel disease. Semin Immunol. 2011 Apr;23(2):130-8. doi: 10.1016/j.smim.2011.01.012. Epub 2011 Feb 3. PMID 21295492
- [Background] Mallone R, Mannering SI, Brooks-Worrell BM, Durinovic-Bello I, Cilio CM, Wong FS, Schloot NC; T-Cell Workshop Committee, Immunology of Diabetes Society. Isolation and preservation of peripheral blood mononuclear cells for analysis of islet antigen-reactive T cell responses: position statement of the T-Cell Workshop Committee of the Immunology of Diabetes Society. Clin Exp Immunol. 2011 Jan;163(1):33-49. doi: 10.1111/j.1365-2249.2010.04272.x. Epub 2010 Oct 5. PMID 20939860
- [Background] Nalleweg N, Chiriac MT, Podstawa E, Lehmann C, Rau TT, Atreya R, Krauss E, Hundorfean G, Fichtner-Feigl S, Hartmann A, Becker C, Mudter J. IL-9 and its receptor are predominantly involved in the pathogenesis of UC. Gut. 2015 May;64(5):743-55. doi: 10.1136/gutjnl-2013-305947. Epub 2014 Jun 23. PMID 24957265
- [Background] Cooper MA, Fehniger TA, Caligiuri MA. The biology of human natural killer-cell subsets. Trends Immunol. 2001 Nov;22(11):633-40. doi: 10.1016/s1471-4906(01)02060-9. PMID 11698225
- [Background] Soler D, Chapman T, Yang LL, Wyant T, Egan R, Fedyk ER. The binding specificity and selective antagonism of vedolizumab, an anti-alpha4beta7 integrin therapeutic antibody in development for inflammatory bowel diseases. J Pharmacol Exp Ther. 2009 Sep;330(3):864-75. doi: 10.1124/jpet.109.153973. Epub 2009 Jun 9. PMID 19509315
- [Background] Iellem A, Colantonio L, D'Ambrosio D. Skin-versus gut-skewed homing receptor expression and intrinsic CCR4 expression on human peripheral blood CD4+CD25+ suppressor T cells. Eur J Immunol. 2003 Jun;33(6):1488-96. doi: 10.1002/eji.200323658. PMID 12778466
- [Background] Li L, Boussiotis VA. Molecular and functional heterogeneity of T regulatory cells. Clin Immunol. 2011 Dec;141(3):244-52. doi: 10.1016/j.clim.2011.08.011. Epub 2011 Aug 30. PMID 21945485
- [Background] Hovhannisyan Z, Treatman J, Littman DR, Mayer L. Characterization of interleukin-17-producing regulatory T cells in inflamed intestinal mucosa from patients with inflammatory bowel diseases. Gastroenterology. 2011 Mar;140(3):957-65. doi: 10.1053/j.gastro.2010.12.002. Epub 2010 Dec 11. PMID 21147109
- [Background] Menning A, Loddenkemper C, Westendorf AM, Szilagyi B, Buer J, Siewert C, Hamann A, Huehn J. Retinoic acid-induced gut tropism improves the protective capacity of Treg in acute but not in chronic gut inflammation. Eur J Immunol. 2010 Sep;40(9):2539-48. doi: 10.1002/eji.200939938. PMID 20690178
- [Background] Abramson O, Qiu S, Erle DJ. Preferential production of interferon-gamma by CD4+ T cells expressing the homing receptor integrin alpha4/beta7. Immunology. 2001 Jun;103(2):155-63. doi: 10.1046/j.0019-2805.2001.01234.x. PMID 11412302
- [Background] El Azreq MA, Boisvert M, Cesaro A, Page N, Loubaki L, Allaeys I, Chakir J, Poubelle PE, Tessier PA, Aoudjit F. alpha2beta1 integrin regulates Th17 cell activity and its neutralization decreases the severity of collagen-induced arthritis. J Immunol. 2013 Dec 15;191(12):5941-50. doi: 10.4049/jimmunol.1301940. Epub 2013 Nov 15. PMID 24244022
- [Background] Baaten BJ, Cooper AM, Swain SL, Bradley LM. Location, location, location: the impact of migratory heterogeneity on T cell function. Front Immunol. 2013 Oct 8;4:311. doi: 10.3389/fimmu.2013.00311. PMID 24115949
- [Background] Munger JS, Huang X, Kawakatsu H, Griffiths MJ, Dalton SL, Wu J, Pittet JF, Kaminski N, Garat C, Matthay MA, Rifkin DB, Sheppard D. The integrin alpha v beta 6 binds and activates latent TGF beta 1: a mechanism for regulating pulmonary inflammation and fibrosis. Cell. 1999 Feb 5;96(3):319-28. doi: 10.1016/s0092-8674(00)80545-0. PMID 10025398
- [Background] Travis MA, Reizis B, Melton AC, Masteller E, Tang Q, Proctor JM, Wang Y, Bernstein X, Huang X, Reichardt LF, Bluestone JA, Sheppard D. Loss of integrin alpha(v)beta8 on dendritic cells causes autoimmunity and colitis in mice. Nature. 2007 Sep 20;449(7160):361-5. doi: 10.1038/nature06110. Epub 2007 Aug 12. PMID 17694047
- [Background] Bridges LC, Sheppard D, Bowditch RD. ADAM disintegrin-like domain recognition by the lymphocyte integrins alpha4beta1 and alpha4beta7. Biochem J. 2005 Apr 1;387(Pt 1):101-8. doi: 10.1042/BJ20041444. PMID 15504110
- [Background] Hynes RO. Integrins: bidirectional, allosteric signaling machines. Cell. 2002 Sep 20;110(6):673-87. doi: 10.1016/s0092-8674(02)00971-6. PMID 12297042
- [Background] Han JM, Patterson SJ, Levings MK. The Role of the PI3K Signaling Pathway in CD4(+) T Cell Differentiation and Function. Front Immunol. 2012 Aug 13;3:245. doi: 10.3389/fimmu.2012.00245. eCollection 2012. PMID 22905034
- [Background] Assi K, Patterson S, Dedhar S, Owen D, Levings M, Salh B. Role of epithelial integrin-linked kinase in promoting intestinal inflammation: effects on CCL2, fibronectin and the T cell repertoire. BMC Immunol. 2011 Aug 1;12:42. doi: 10.1186/1471-2172-12-42. PMID 21806815
- [Background] Schiering C, Krausgruber T, Chomka A, Frohlich A, Adelmann K, Wohlfert EA, Pott J, Griseri T, Bollrath J, Hegazy AN, Harrison OJ, Owens BMJ, Lohning M, Belkaid Y, Fallon PG, Powrie F. The alarmin IL-33 promotes regulatory T-cell function in the intestine. Nature. 2014 Sep 25;513(7519):564-568. doi: 10.1038/nature13577. Epub 2014 Jul 16. PMID 25043027
- [Background] Cohen CJ, Crome SQ, MacDonald KG, Dai EL, Mager DL, Levings MK. Human Th1 and Th17 cells exhibit epigenetic stability at signature cytokine and transcription factor loci. J Immunol. 2011 Dec 1;187(11):5615-26. doi: 10.4049/jimmunol.1101058. Epub 2011 Nov 2. PMID 22048764
- [Background] Iwata M, Hirakiyama A, Eshima Y, Kagechika H, Kato C, Song SY. Retinoic acid imprints gut-homing specificity on T cells. Immunity. 2004 Oct;21(4):527-38. doi: 10.1016/j.immuni.2004.08.011. PMID 15485630
- [Background] Bakdash G, Vogelpoel LT, van Capel TM, Kapsenberg ML, de Jong EC. Retinoic acid primes human dendritic cells to induce gut-homing, IL-10-producing regulatory T cells. Mucosal Immunol. 2015 Mar;8(2):265-78. doi: 10.1038/mi.2014.64. Epub 2014 Jul 16. PMID 25027601
- [Background] Kempster SL, Kaser A. alpha4beta7 integrin: beyond T cell trafficking. Gut. 2014 Sep;63(9):1377-9. doi: 10.1136/gutjnl-2013-305967. Epub 2013 Dec 11. No abstract available. PMID 24334217
- [Background] Denucci CC, Mitchell JS, Shimizu Y. Integrin function in T-cell homing to lymphoid and nonlymphoid sites: getting there and staying there. Crit Rev Immunol. 2009;29(2):87-109. doi: 10.1615/critrevimmunol.v29.i2.10. PMID 19496742
- [Background] Teague TK, Lazarovits AI, McIntyre BW. Integrin alpha 4 beta 7 co-stimulation of human peripheral blood T cell proliferation. Cell Adhes Commun. 1994 Dec;2(6):539-47. doi: 10.3109/15419069409014217. PMID 7743139
- [Background] Briskin M, Winsor-Hines D, Shyjan A, Cochran N, Bloom S, Wilson J, McEvoy LM, Butcher EC, Kassam N, Mackay CR, Newman W, Ringler DJ. Human mucosal addressin cell adhesion molecule-1 is preferentially expressed in intestinal tract and associated lymphoid tissue. Am J Pathol. 1997 Jul;151(1):97-110. PMID 9212736
- [Background] Souza HS, Elia CC, Spencer J, MacDonald TT. Expression of lymphocyte-endothelial receptor-ligand pairs, alpha4beta7/MAdCAM-1 and OX40/OX40 ligand in the colon and jejunum of patients with inflammatory bowel disease. Gut. 1999 Dec;45(6):856-63. doi: 10.1136/gut.45.6.856. PMID 10562584
- [Background] Himmel ME, MacDonald KG, Garcia RV, Steiner TS, Levings MK. Helios+ and Helios- cells coexist within the natural FOXP3+ T regulatory cell subset in humans. J Immunol. 2013 Mar 1;190(5):2001-8. doi: 10.4049/jimmunol.1201379. Epub 2013 Jan 28. PMID 23359504
- [Background] McMurchy AN, Levings MK. Suppression assays with human T regulatory cells: a technical guide. Eur J Immunol. 2012 Jan;42(1):27-34. doi: 10.1002/eji.201141651. Epub 2011 Dec 12. PMID 22161814
- [Background] Wu X, Lahiri A, Haines GK 3rd, Flavell RA, Abraham C. NOD2 regulates CXCR3-dependent CD8+ T cell accumulation in intestinal tissues with acute injury. J Immunol. 2014 Apr 1;192(7):3409-18. doi: 10.4049/jimmunol.1302436. Epub 2014 Mar 3. PMID 24591373
- [Background] Ramesh G, Alvarez X, Borda JT, Aye PP, Lackner AA, Sestak K. Visualizing cytokine-secreting cells in situ in the rhesus macaque model of chronic gut inflammation. Clin Diagn Lab Immunol. 2005 Jan;12(1):192-7. doi: 10.1128/CDLI.12.1.192-197.2005. PMID 15643006